CLINICAL TRIAL: NCT02487030
Title: A Phase 3, Randomized, Open-Label, Study to Evaluate the Safety and Efficacy of Ledipasvir/Sofosbuvir Fixed Dose Combination, With or Without Ribavirin, in Egyptian Adults With Chronic Genotype 4 HCV Infection
Brief Title: Safety and Efficacy of Ledipasvir/Sofosbuvir Fixed Dose Combination, With or Without Ribavirin, in Egyptian Adults With Chronic Genotype 4 HCV Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-337-1643
Record Dates: First submitted 2015-06-27; First posted 2015-07-01 (Estimated); Results first posted 2017-12-14 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2017-11

CONDITIONS: Hepatitis C Virus Infection
Keywords: HCV genotype 4 (GT-4); HCV; Sustained Virologic Response; Direct Acting Antiviral; Combination Therapy; GS-7977; GS-5885; Ribavirin; Sofosbuvir; ledipasvir; Hepatitis C; Hepatitis C, Chronic; Liver Diseases; Virus Diseases; Antiviral Agents
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic; Liver Diseases; Virus Diseases | interventions — ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (7):
- LDV/SOF 8 wk TN (Cohort 1, Group 1) (Experimental): LDV/SOF for 8 weeks (treatment-naive (TN))
  Interventions: Drug: LDV/SOF
- LDV/SOF+RBV 8 wk TN (Cohort 1, Group 2) (Experimental): LDV/SOF+RBV for 8 weeks (treatment-naive)
  Interventions: Drug: LDV/SOF; Drug: RBV
- LDV/SOF 12 wk TN (Cohort 1, Group 3) (Experimental): LDV/SOF for 12 weeks (treatment-naive)
  Interventions: Drug: LDV/SOF
- LDV/SOF+RBV 12 wk TN (Cohort 1, Group 4) (Experimental): LDV/SOF+RBV for 12 weeks (treatment-naive)
  Interventions: Drug: LDV/SOF; Drug: RBV
- LDV/SOF+RBV 12 wk TE (Cohort 2) (Experimental): Treatment-experienced (TE) participants who completed treatment in Gilead sponsored study GS-US-334-0138 or in Cohort 1 of this study and did not achieve SVR12 will receive LDV/SOF+RBV for 12 weeks.
  Interventions: Drug: LDV/SOF; Drug: RBV
- LDV/SOF 12 wk TE (Cohort 3, Group 1) (Experimental): LDV/SOF for 12 weeks (treatment-experienced)
  Interventions: Drug: LDV/SOF
- LDV/SOF+RBV 12 wk TE (Cohort 3, Group 2) (Experimental): LDV/SOF+RBV for 12 weeks (treatment-experienced)
  Interventions: Drug: LDV/SOF; Drug: RBV

INTERVENTIONS:
Drug: LDV/SOF — 90/400 mg FDC tablet administered orally once daily
  Other Names: Harvoni®; GS-5885/GS-7977
Drug: RBV — Tablets administered orally in a divided daily dose based on weight (< 75 kg = 1000 mg and ≥ 75 kg = 1200 mg)
  Arms: LDV/SOF+RBV 12 wk TE (Cohort 2); LDV/SOF+RBV 12 wk TE (Cohort 3, Group 2); LDV/SOF+RBV 12 wk TN (Cohort 1, Group 4); LDV/SOF+RBV 8 wk TN (Cohort 1, Group 2)

SUMMARY:
The primary objective of this study was to evaluate the efficacy, safety, and tolerability of ledipasvir/sofosbuvir (LDV/SOF) fixed dose combination (FDC) with or without ribavirin (RBV) in Egyptian adults with chronic genotype 4 hepatitis C virus (HCV) infection.

ELIGIBILITY:
Key Inclusion Criteria:

* Willing and able to provide written informed consent
* Chronic HCV infection (≥ 6 months) documented by medical history or liver biopsy
* HCV genotype 4 at screening
* HCV treatment naive or prior participation in this study or study GS-US-334-0138 (Cohorts 1 and 2 only)
* Cohort 3 only: HCV treatment-experienced (previously received therapy for HCV infection with an interferon (IFN)-containing regimen, with or without RBV and/or an HCV NS3/NS4A protease inhibitor (PI)
* Body mass index (BMI) ≥ 18 kg/m^2
* Screening laboratory values within defined thresholds
* Use of effective protocol-approved contraception methods

Key Exclusion Criteria:

* History of clinically-significant illness or any other major medical disorder that may interfere with treatment, assessment or compliance with the protocol
* Infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV)
* Pregnant or nursing females or male with pregnant female partner
* Clinically-relevant drug or alcohol abuse within 12 months of screening

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2015-09-07 (Actual); Primary Completion 2016-11-11 (Actual); Study Completion 2017-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (3):
- Egypt (3):
  - Al Mansurah
  - Cairo
  - Shibīn al Kawm

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Result] Shiha G, Waked I, Soliman R, Abdelrazek W, Hassany M, Fouad R, et al. Ledipasvir/sofosbuvir for 8 or 12 weeks with or without ribavirin in HCV genotype 4 patients in Egypt. [Abstract OP158]. Asian Pacific Association for the Study of the Liver (APASL); 2017 15-19 February; Shanghai, China
- [Derived] Shiha G, Esmat G, Hassany M, Soliman R, Elbasiony M, Fouad R, Elsharkawy A, Hammad R, Abdel-Razek W, Zakareya T, Kersey K, Massetto B, Osinusi A, Lu S, Brainard DM, McHutchison JG, Waked I, Doss W. Ledipasvir/sofosbuvir with or without ribavirin for 8 or 12 weeks for the treatment of HCV genotype 4 infection: results from a randomised phase III study in Egypt. Gut. 2019 Apr;68(4):721-728. doi: 10.1136/gutjnl-2017-315906. Epub 2018 Apr 17. PMID 29666174

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in 4 sites in Egypt. The first participant was screened on 07 September 2015 and the last study visit was on 04 February 2017.
Pre-assignment Details: 289 participants were screened.
Groups:
- LDV/SOF 8 wk TN (Cohort 1, Group 1): Ledipasvir/sofosbuvir (Harvoni®; LDV/SOF) (90/400 mg) fixed dose combination (FDC) tablet administered orally once daily for 8 weeks (wk) in treatment-naive (TN) participants
- LDV/SOF + RBV 8 wk TN (Cohort 1, Group 2): LDV/SOF (90/400 mg) FDC tablet administered orally once daily + Ribavirin (RBV) tablets administered orally in a divided daily dose based on weight (< 75 kg = 1000 mg and ≥ 75 kg = 1200 mg) for 8 weeks in TN participants
- LDV/SOF 12 wk TN (Cohort 1, Group 3): LDV/SOF (90/400 mg) FDC tablet administered orally once daily for 12 weeks in TN participants
- LDV/SOF + RBV 12 wk TN (Cohort 1, Group 4): LDV/SOF (90/400 mg) FDC tablet administered orally once daily + RBV tablets administered orally in a divided daily dose based on weight (< 75 kg = 1000 mg and ≥ 75 kg = 1200 mg) for 12 weeks in TN participants
- LDV/SOF 12 wk TE (Cohort 3, Group 1): LDV/SOF (90/400 mg) FDC tablet administered orally once daily in treatment-experienced (TE) participants
- LDV/SOF + RBV 12 wk TE (Cohort 3, Group 2): LDV/SOF (90/400 mg) FDC tablet administered orally once daily + RBV tablets administered orally in a divided daily dose based on weight (< 75 kg = 1000 mg and ≥ 75 kg = 1200 mg) for 12 weeks in TE participants
- LDV/SOF + RBV 12 wk SOF or LDV/SOF Experienced (Cohort 2): LDV/SOF (90/400 mg) FDC tablet administered orally once daily + RBV tablets administered orally in a divided daily dose based on weight (< 75 kg = 1000 mg and ≥ 75 kg = 1200 mg) for 12 weeks in SOF or LDV/SOF experienced participants. Participants who completed treatment in Study GS-US-334-0138 with SOF+RBV for 12 or 24 weeks or those who participated in Cohort 1 of this study with LDV/SOF ± RBV for 8 weeks and did not achieve SVR12 were in enrolled into Cohort 2.
Period: Overall Study
Arm/Group | LDV/SOF 8 wk TN (Cohort 1, Group 1) | LDV/SOF + RBV 8 wk TN (Cohort 1, Group 2) | LDV/SOF 12 wk TN (Cohort 1, Group 3) | LDV/SOF + RBV 12 wk TN (Cohort 1, Group 4) | LDV/SOF 12 wk TE (Cohort 3, Group 1) | LDV/SOF + RBV 12 wk TE (Cohort 3, Group 2) | LDV/SOF + RBV 12 wk SOF or LDV/SOF Experienced (Cohort 2)
Started | 43 | 42 | 43 | 42 | 36 | 38 | 11
Completed | 41 | 38 | 41 | 40 | 34 | 37 | 11
Not Completed | 2 | 4 | 2 | 2 | 2 | 1 | 0
Not completed — Lack of Efficacy | 2 | 4 | 1 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who were randomized or enrolled and received at least 1 dose of study drug
Groups:
- LDV/SOF 8 wk TN (Cohort 1, Group 1): LDV/SOF (90/400 mg) FDC tablet administered orally once daily for 8 weeks in TN participants
- LDV/SOF + RBV 8 wk TN (Cohort 1, Group 2): LDV/SOF (90/400 mg) FDC tablet administered orally once daily + RBV tablets administered orally in a divided daily dose based on weight (< 75 kg = 1000 mg and ≥ 75 kg = 1200 mg) for 8 weeks in TN participants
- LDV/SOF 12 wk TE (Cohort 3, Group 1): LDV/SOF (90/400 mg) FDC tablet administered orally once daily in TE participants
- LDV/SOF + RBV 12 wk SOF or LDV/SOF Experienced (Cohort 2): LDV/SOF (90/400 mg) FDC tablet administered orally once daily + RBV tablets administered orally in a divided daily dose based on weight (< 75 kg = 1000 mg and ≥ 75 kg = 1200 mg) for 12 weeks in SOF or LDV/SOF experienced participants. Participants who completed treatment in Study GS-US-334-0138 with SOF+RBV for 12 or 24 weeks or those who participated in Cohort 1 of this study with LDV/SOF ± RBV for 8 weeks and did not achieve SVR12 were enrolled into Cohort 2.
- Total: Total of all reporting groups
Arm/Group | LDV/SOF 8 wk TN (Cohort 1, Group 1) | LDV/SOF + RBV 8 wk TN (Cohort 1, Group 2) | LDV/SOF 12 wk TN (Cohort 1, Group 3) | LDV/SOF + RBV 12 wk TN (Cohort 1, Group 4) | LDV/SOF 12 wk TE (Cohort 3, Group 1) | LDV/SOF + RBV 12 wk TE (Cohort 3, Group 2) | LDV/SOF + RBV 12 wk SOF or LDV/SOF Experienced (Cohort 2) | Total
Number analyzed (Participants) | 43 | 42 | 43 | 42 | 36 | 38 | 11 | 255
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (13.9) | 49 (12.2) | 49 (13.0) | 46 (12.1) | 49 (11.8) | 51 (10.1) | 48 (16.3) | 50.0 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 21 | 20 | 4 | 13 | 3 | 99
  Male | 25 | 22 | 22 | 22 | 32 | 25 | 8 | 156
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 43 | 42 | 43 | 42 | 36 | 38 | 11 | 255
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 43 | 42 | 43 | 42 | 36 | 38 | 11 | 255
IL28b Status [Count of Participants; unit: Participants] — The CC, CT, and TT alleles are different forms of the IL28b gene.
  Participants
    CC | 12 | 5 | 11 | 9 | 8 | 8 | 0 | 53
    CT | 28 | 26 | 26 | 25 | 24 | 21 | 8 | 158
    TT | 3 | 11 | 6 | 8 | 7 | 9 | 3 | 47
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL)] | 6.0 (0.64) | 5.6 (0.63) | 5.7 (0.69) | 5.8 (0.66) | 5.8 (1.10) | 5.8 (1.04) | 6.2 (0.59) | 5.8 (0.79)
HCV RNA Category [Count of Participants; unit: Participants]
  < 800,000 IU/mL | 17 | 26 | 25 | 28 | 16 | 17 | 5 | 134
  ≥ 800,000 IU/mL | 26 | 16 | 18 | 14 | 20 | 21 | 6 | 121

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ) 12 weeks following the last dose of study drug.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: all randomized or enrolled participants who had genotype 4 HCV infection and who took at least 1 dose of study drug.
Measure: Number (99% Confidence Interval); unit: percentage of participants
Arm/Group | LDV/SOF 8 wk TN (Cohort 1, Group 1) | LDV/SOF + RBV 8 wk TN (Cohort 1, Group 2) | LDV/SOF 12 wk TN (Cohort 1, Group 3) | LDV/SOF + RBV 12 wk TN (Cohort 1, Group 4) | LDV/SOF 12 wk TE (Cohort 3, Group 1) | LDV/SOF + RBV 12 wk TE (Cohort 3, Group 2) | LDV/SOF + RBV 12 wk SOF or LDV/SOF Experienced (Cohort 2)
Number analyzed (Participants) | 43 | 42 | 43 | 42 | 36 | 38 | 11
percentage of participants | 95.3 [84.2 to 99.4] | 90.5 [77.4 to 97.3] | 97.7 [87.7 to 99.9] | 97.6 [87.4 to 99.9] | 94.4 [81.3 to 99.3] | 100.0 [90.7 to 100.0] | 100.0 [71.5 to 100.0]

2. Primary Outcome: Percentage of Participants Who Discontinued LDV/SOF Drug Due to an Adverse Event (AE)
Time Frame: 12 weeks
Population: Safety analysis Set
Measure: Number; unit: percentage of participants
Groups:
- LDV/SOF 8 Weeks: LDV/SOF (90/400 mg) FDC tablet administered orally once daily for 8 weeks
- LDV/SOF + RBV 8 Weeks; LDV/SOF + RBV 12 Weeks: LDV/SOF (90/400 mg) FDC tablet administered orally once daily + RBV tablets administered orally in a divided daily dose based on weight (< 75 kg = 1000 mg and ≥ 75 kg = 1200 mg) for 8 weeks
- LDV/SOF 12 Weeks: LDV/SOF (90/400 mg) FDC tablet administered orally once daily for 12 weeks
Arm/Group | LDV/SOF 8 Weeks | LDV/SOF + RBV 8 Weeks | LDV/SOF 12 Weeks | LDV/SOF + RBV 12 Weeks
Number analyzed (Participants) | 43 | 42 | 79 | 91
percentage of participants | 0 | 0 | 0 | 1.1

3. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 4 and 24 Weeks After Discontinuation of Therapy (SVR4 and SVR24)
Description: SVR4 and SVR24 were defined as HCV RNA < LLOQ 4 and 24 weeks after the last dose of study drug, respectively.
Time Frame: Posttreatment Weeks 4 and 24
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LDV/SOF 8 wk TN (Cohort 1, Group 1) | LDV/SOF + RBV 8 wk TN (Cohort 1, Group 2) | LDV/SOF 12 wk TN (Cohort 1, Group 3) | LDV/SOF + RBV 12 wk TN (Cohort 1, Group 4) | LDV/SOF 12 wk TE (Cohort 3, Group 1) | LDV/SOF + RBV 12 wk TE (Cohort 3, Group 2) | LDV/SOF + RBV 12 wk SOF or LDV/SOF Experienced (Cohort 2)
Number analyzed (Participants) | 43 | 42 | 43 | 42 | 36 | 38 | 11
percentage of participants
  SVR4 | 95.3 [84.2 to 99.4] | 95.2 [83.8 to 99.4] | 97.7 [87.7 to 99.9] | 97.6 [87.4 to 99.9] | 100.0 [90.3 to 100.0] | 100.0 [90.7 to 100.0] | 100.0 [71.5 to 100.0]
  SVR24 | 95.3 [84.2 to 99.4] | 90.5 [77.4 to 97.3] | 97.7 [87.7 to 99.9] | 97.6 [87.4 to 99.9] | 94.4 [81.3 to 99.3] | 100.0 [90.7 to 100.0] | 100.0 [71.5 to 100.0]

4. Secondary Outcome: Percentage of Participants With Overall Virologic Failure
Description: Virologic failure was defined as
  * On-treatment virologic failure
    * confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ, while on treatment (ie, breakthrough),
    * confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment (ie, rebound),
    * HCV RNA persistently ≥ LLOQ through 8 weeks of treatment (ie, nonresponse)
  * Relapse
    * HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at end of treatment, confirmed with 2 consecutive values or last available posttreatment measurement
Time Frame: Up to Posttreatment Week 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 8 wk TN (Cohort 1, Group 1) | LDV/SOF + RBV 8 wk TN (Cohort 1, Group 2) | LDV/SOF 12 wk TN (Cohort 1, Group 3) | LDV/SOF + RBV 12 wk TN (Cohort 1, Group 4) | LDV/SOF 12 wk TE (Cohort 3, Group 1) | LDV/SOF + RBV 12 wk TE (Cohort 3, Group 2) | LDV/SOF + RBV 12 wk SOF or LDV/SOF Experienced (Cohort 2)
Number analyzed (Participants) | 43 | 42 | 43 | 42 | 36 | 38 | 11
percentage of participants | 4.7 | 9.5 | 2.3 | 0.0 | 2.8 | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: Up to 12 weeks + 30 days
Arm/Group | LDV/SOF 8 Weeks | LDV/SOF + RBV 8 Weeks | LDV/SOF 12 Weeks | LDV/SOF + RBV 12 Weeks
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/42 | 0/79 | 3/91
Other Adverse Events (participants affected / at risk) | 11/43 | 15/42 | 23/79 | 41/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF 8 Weeks (N=43) | LDV/SOF + RBV 8 Weeks (N=42) | LDV/SOF 12 Weeks (N=79) | LDV/SOF + RBV 12 Weeks (N=91)
Chest Pain (General disorders) | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF 8 Weeks (N=43) | LDV/SOF + RBV 8 Weeks (N=42) | LDV/SOF 12 Weeks (N=79) | LDV/SOF + RBV 12 Weeks (N=91)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 7
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 0 | 6
Constipation (Gastrointestinal disorders) | 0 | 3 | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 3 | 1 | 5 | 6
Fatigue (General disorders) | 4 | 5 | 8 | 14
Pyrexia (General disorders) | 1 | 1 | 1 | 5
Bronchitis (Infections and infestations) | 3 | 1 | 3 | 2
Headache (Nervous system disorders) | 4 | 13 | 13 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years